CLINICAL TRIAL: NCT07176910
Title: Doppler Ultrasound-Guided Angiopuncture for Dysmenorrhea Pain: A Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Collaborators: The Third Affiliated Hospital of Changchun University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Rong Han, PhD student, City University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111; 9239056 (Other Grant/Funding Number: This study was supported by Health Evaluation and Intervention Using Advanced Raymedy System of Raymedy Bio-Energy Inn)
Record Dates: First submitted 2025-09-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Angiopuncture; Dysmenorrhea; Dopplar Ultrasound
Keywords: Dysmenorrhea; angiopuncture; dopplar; ultrasound
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: unmarried nulliparous women (aged 18-25 years old) with dysmenorrhea diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- angiopuncture treated group (Experimental): conduct angiopuncture therapy
  Interventions: Other: conduct angiopuncture on perforator points

INTERVENTIONS:
Other: conduct angiopuncture on perforator points — conducted angiopuncutre on patients of intervention group, and compare those patients pain scores before and after angiopuncture therapy.

SUMMARY:
the study is to evaluated dopplar guided angiopuncture efficacy and safety in patients with dysmenorrhea

DETAILED DESCRIPTION:
to conduct angiopuncture, with dopplar located perforator points and also evaluate the spectrum before and after angiopuncture therapy.

ELIGIBILITY:
Inclusion Criteria:

Primary dysmenorrhea diagnosis (≥6 months of menstrual pain scoring ≥2 on numerical rating scale) Regular menstrual cycles (28-32 days), menstrual period lasts 4 to 7 days No pelvic pathology on transvaginal ultrasound.

Exclusion Criteria:

coagulopathy (INR >1.5) recent analgesic use (48-hour washout) secondary dysmenorrhea confirmed by laparoscopy.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since we studied dysmenorrhea, we recuited nmarried nulliparous women.
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale | pre-treatment, immediate post-treatment, check up 1, check up 2, check up 3 (3 check ups lasts for 3 months post therapy, with each for 1 month)
  to measure pain score before and after angiopuncture

CONTACTS AND LOCATIONS:
Overall Officials: Jinlian HU, PhD, Principal Investigator — City University of Hong Kong
Locations (1):
- The Third Affiliated Hospital of Changchun University of Chinese Medicine, Changchun, China

IPD SHARING:
Plan to Share IPD: No
we have not published the paper yet